CLINICAL TRIAL: NCT04473235
Title: Better Memory With Literacy Acquisition Later in Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Federal University of Minas Gerais (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P0541386; R21AG069252 (NIH)
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Memory Impairment
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Literacy training (Experimental): The basic-literacy training will be given for two hours/day for four days/week for 6 months. At baseline, participants will be randomized into four classes of 30. An expert in adult education will oversee the classes and meet the teachers periodically, and each class will count with a certified and experienced lead teacher and teacher aid. The intervention group will receive literacy training based on analytical and phonemic methods for enabling reading and writing
  Interventions: Behavioral: Literacy training
- Non-literacy training (Active Comparator): The comparator group will have access to non-literacy classes offered at the adult school, including geography, history, informatics, and sciences, but no literacy-training, for two hours/day for four days/week for 6 months.
  Interventions: Behavioral: Non-Literacy training

INTERVENTIONS:
Behavioral: Literacy training — Teaching adults how to read and write using the analytical and phonemic method
  Arms: Literacy training
Behavioral: Non-Literacy training — Attending classes in geography, history, sciences, without receiving the specific training in literacy
  Arms: Non-literacy training

SUMMARY:
This study aims to discover whether acquiring basic-literacy in adulthood can improve episodic memory and brain structural and functional connectivity. In a collaborative project between Brazil and USA, the investigators will use a randomized controlled trial approach to leverage the level of evidence of the benefits of basic adult-education as a possible cognitive reserve builder. If successful, the study's findings will be important in shaping policies targeting increasing access to late-life education to reduce dementia risk.

ELIGIBILITY:
Inclusion Criteria:

Being illiterate (TOFHLA score <53) and availability to participate in the study for at least 12 months

Exclusion Criteria:

A) Presence of remarkable cognitive complains and/or decompensated psychiatric illness (depression and anxiety) and/or current substance abuse such as alcohol and illicit drugs use.

B) Objective cognitive impairment: score of 2 standard deviations or bellow for age and education on the Mini-Mental State Evaluation (MMSE) and/or score of 6 or lower on the delayed recall task from the Brief Cognitive Battery.

C) History of previously diagnosed dyslexia D) Formal MRI contraindications including metal or claustrophobia. E) Severe structural lesions detected by MRI.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Resende, MD, PhD, Principal Investigator — UFMG; Lea T Grinberg, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The assignment of participants to each arm group occured after enrollment. There was no specific event before assigment.
Period: Overall Study
Arm/Group | Literacy Training | Non-literacy Training
Started | 58 | 50
Completed | 39 | 38
Not Completed | 19 | 12
Not completed — Lost to Follow-up | 6 | 5
Not completed — Declined continuation | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Literacy Training | Non-literacy Training | Total
Number analyzed (Participants) | 58 | 50 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.8) | 58.4 (9.7) | 58.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 77
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 50 | 108
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 39 | 78
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 7 | 21
Region of Enrollment [Number; unit: participants]
  Brazil | 58 | 50 | 108
Free and cued recall sum of attempts [Mean (Standard Deviation); unit: units on a scale] — The Free and Cued Selective Reminding Test (FCSRT) is an episodic memory test. First, the participant learns 16 figures, 4 each time, with the help of semantic cues provided by the examiner. After that, the participant recalls the figures 3 times, with a distraction activity between each attempt (counting 20 to 1 backwards). The sum of each immediate free recall is called sum of attempts. It ranges from 0 (the participant does not recall any figure in three attempts) to 48 (the participant recalls all the figures). The higher the score, the better the participant's episodic memory.
  units on a scale | 28.3 (7.1) | 28.4 (5.5) | 28.3 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Episodic Memory Improvement
Description: Change in free recall sum-of-attempts of the Free and Cued Selective Reminding with Immediate Recall (FCSR) test.
  The Free and Cued Selective Reminding Test (FCSRT) is an episodic memory test. First, the participant learns 16 figures, 4 each time, with the help of semantic cues provided by the examiner. After that, the participant recalls the figures 3 times, with a distraction activity between each attempt (counting 20 to 1 backwards). The sum of each immediate free recall is called sum of attempts. It ranges from 0 (the participant does not recall any figure in three attempts) to 48 (the participant recalls all the figures). The higher the score, the better the participant's episodic memory.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Literacy Training | Non-literacy Training
Number analyzed (Participants) | 39 | 38
score on a scale | 31.8 (5.8) | 31.3 (5.5)
Statistical Analysis 1: Comparison: Literacy Training vs Non-literacy Training; Test type: Superiority; p = 0.531, t-test, 2 sided; Mean Difference (Final Values) = -0.799, Standard Error of Mean 1.3

2. Secondary Outcome: Change in Brain Connectivity
Description: The intrinsic functional connectivity will be measured using the BOLD (blood oxygen level dependent) that is calculated through resting state functional MRIs that will be performed at baseline and at 6 months follow up. After preprocessing the images and accounting for potential cofounders (head motion signal, cerebral spinal signal, physiological signal and white matter signal), the BOLD signal is measured and coregistered in T1 images for anatomical correspondence of the signal. Then, a seed is placed in the hippocampus and the BOLD signal between the hippocampus and the prefrontal cortex is calculated at baseline and at 6 months follow up. The higher the value, the more the regions are connected. Change in the intrinsic functional connectivity between the hippocampus and the prefrontal cortex.
Time Frame: Baseline and 6 months
Population: Some participants had artifacts in their MRIs that made the researchers not able to interpret the resting state functional MRI. Therefore these participants are not included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Literacy Training | Non-literacy Training
Number analyzed (Participants) | 31 | 32
unitless
  Connectivity between the left hippocampal and left prefrontal cortex | -0.11 (0.38) | 0.06 (0.39)
  Connectivity between the right hippocampal and right prefrontal cortex | -0.11 (0.42) | -0.05 (0.39)
Statistical Analysis 1: Comparison: Literacy Training vs Non-literacy Training; Difference in the connectivity between the left hippocampus and left prefrontal cortex; Test type: Superiority; p = 0.627, t-test, 2 sided; Mean Difference (Final Values) = 0.02
Statistical Analysis 2: Comparison: Literacy Training vs Non-literacy Training; Difference in the connectivity between the right hippocampus and right prefrontal cortex; Test type: Superiority; p = 0.120, t-test, 2 sided; Mean Difference (Final Values) = 0.08

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Non-literacy Training: The comparator group will have access to non-literacy classes offered at the adult school, including geography, history, informatics, and sciences, but no literacy-training, for two hours/day for four days/week for 6 months. After 6 months, the groups switch, so the comparator receives the specific reading and writing training, and the intervention group receives the lessons on other themes.
  Non-Literacy training: Attending classes in geography, history, sciences, without receiving the specific training in literacy
Arm/Group | Literacy Training | Non-literacy Training
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/50
Other Adverse Events (participants affected / at risk) | 1/58 | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Literacy Training (N=58) | Non-literacy Training (N=50)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Claustrofobia (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04473235/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT04473235/SAP_001.pdf
  • Informed Consent Form (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04473235/ICF_002.pdf